CLINICAL TRIAL: NCT06785480
Title: Evaluation of Computer-controlled Local Anesthesia in Children - a Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC-09243
Record Dates: First submitted 2025-01-09; First posted 2025-01-21 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Local Anesthesia Injection Pain
Keywords: dentistry; pediatric; local anesthesia; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Split Mouth Design In this randomized controlled study, each patient undergoes two separate dental treatments, bilateral in the upper jaw. Each patient will receive local anesthesia once administered using the CCLAD device and another time using the conventional syringe. There is at least on week in between the two treatments. This study design effectively employs each patient as their own control, allowing for a direct within-person comparison of the two anesthesia delivery methods The participants are randomized through block randomization for type of local anesthesia and starting side of the mouth (left or right).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CCLAD (Experimental): The CCLAD device is used to administers local anesthesia with 1.2ml Septanest normal (4% articaine, 1/200000 adrenaline). It is set to 60sec/ml in continuous mode. All participants receive this intervention on one randomly assigned side of the mouth.
  Interventions: Device: Computer Controlled Local Anesthetic Delivery (CCLAD)
- Conventional syringe (Active Comparator): A conventional metallic syringe is used to administers local anesthesia with 1.2ml Septanest normal (4% articaine, 1/200000 adrenaline). All participants receive this intervention on one randomly assigned side of the mouth.
  Interventions: Device: Conventional metallic syringe

INTERVENTIONS:
Device: Computer Controlled Local Anesthetic Delivery (CCLAD) — Administering local anesthesia with 1.2ml Septanest normal (4% articaine, 1/200000 adrenaline) with CCLAD. The CCLAD device is set to 60sec/ml in continuous mode.
  Arms: CCLAD
Device: Conventional metallic syringe — A conventional metallic syringe is used to administers local anesthesia with 1.2ml Septanest normal (4% articaine, 1/200000 adrenaline).
  Arms: Conventional syringe

SUMMARY:
The goal of this clinical trial is to learn if Computer Controlled Local Anesthetic Delivery (CCLAD) results in lower pain during local anesthesia administration for infiltration in the buccal region of the upper jaw in patients between 6 and 16 years old who will receive a dental treatment.

The main questions it aims to answer are:

* Does CCLAD result in lower self-reported pain (Visual Analogue Scale (VAS) and Face Pain Scale-Revised (FPS-R)) for patients between 6 and 16 years old who need local anesthesia in the upper jaw for a dental treatment?
* Does CCLADD result in lower observed pain (Sound Eye Motor Scale (SEM)) for patients between 6 and 16 years old who need local anesthesia in the upper jaw for a dental treatment?
* Does CCLAD result in lower hearth rate (HR) and galvanic skin response (GSR) for patients between 6 and 16 years old who need local anesthesia in the upper jaw for a dental treatment? Researchers will compare CCLAD (Dentapen, Septodont, France) to conventional local anesthesia infiltration with a metallic syringe to see if the infiltration is less painful in patients between 6 and 16 years old who will receive a dental treatment.

Participants will receive local anesthesia either with the Dentapen or metallic syringe.

* GSR and heart rate are measured before anesthesia, during needle insertion, at 0.3 - 0.6 - 0.9ml, and after anesthesia.
* Post-injection, the child provides VAS scores (if 8 years or older) and FPS-R (all patients).
* A researcher not administering the injection determines the SEM score.

ELIGIBILITY:
Inclusion criteria:

* Patients between the ages of 6 and 16 years
* Requiring a buccal injection with local anesthesia for dental treatment, bilaterally in the upper jaw
* Treatments: restorative filing, pulpotomy, extraction or a steel crown placement
* At least one week between both treatments
* Complying with the criteria of ASA I (ASA classification of The American Society of Anaesthesiologists, 1963)
* Fluent in Dutch
* Children who had a score of 3 or higher on the Frankl scale

Exclusion criteria:

* Contraindications to inject Local anesthesia (allergy to the liquid, ...)
* Patients referred because of needle phobia or behavior management problems
* Refusing to sign the informed consent

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Immediately after intervention, the child provides VAS scores.
  The Visual Analog Scale is a self-report pain assessment tool applicable from the age of eight. The scale is a 100mm line, where 'no pain' is on the left and 'severe pain' is on the right. Patients indicate the level of pain experienced during local anesthesia by marking this scale. The scale is generally interpretted as follows: 0-4 mm (0-0.4): No pain or mild pain; 5-44 mm (0.5-4.4): Mild pain; 45-74 mm (4.5-7.4): Moderate pain; 75-100 mm (7.5-10): Severe pain. A higher score thus means a worse outcome.
Face Pain Scale-Revised (FPS-R) | Immediately after intervention, the child provides FPS-R scores.
  The Face Pain Scale-Revised (FPS-R) is a self-report pain measurement tool. The scale consists of six gender neutral faces devoid of smiles or tears. Each face corresponds to a score ranging from zero to ten, with only the even numbers used. It is important to employ appropriate language while utilizing the FPS-R. You can use short phrases like 'this face means no pain' or 'this face means very much pain', avoiding the terms 'happy' and 'sad'. In this study the Face Pain Scale-Revised will be used from the age of six. The specific scores for each face from left to right are: 0, 2, 4, 6, 8, 10. A higher score means a worse outcome.

SECONDARY OUTCOMES:
Galvanic Skin Response (GSR) | GSR is measured pre-intervention; periprocedurally during needle insertion at 0.3 - 0.6 - 0.9ml, and immediately after intervention.
  The Galvanic Skin Response, also known as the psychogalvanic Reflex, is used to measure the stress reaction. During local anesthesia, individuals commonly undergo a stress response, triggering an elevation in sympathetic activity. The rise in sympathetic tone activates the sweat glands. As a result, the resistance of the skin decreases, and the electrical conduction increases. To measure these changes, two electrodes are placed, one on the index finger and the other on the middle finger, and these are linked to the application "Mindfield eSense". A higher Galvanic Skin Response is correlated to higher stress and thus a worse outcome.
Heart rate (HR) | Heart rate is measured pre-intervention; periprocedurally during needle insertion at 0.3 - 0.6 - 0.9ml, and immediately after intervention.
  Stress and anxiety trigger the autonomic nervous system. This acts on the parasympathetic system, which is suppressed, and the sympathetic system, which is activated. Due to activation of the sympathetic system epinephrine and norepinephrine are released from the adrenal glands. The release of these hormones causes vasoconstriction in the blood vessels, increased blood pressure and increased heart rate. In this study, the heart rate will be measured with a pulse oximeter. A higher heart rate is a worse outcome.
Sound Eye Motor Scale (SEM) | A researcher not administering the injection determines the SEM score periprocedurally, from the start of injection until 1,2 minutes later when the injection has been completed.
  The Sound Eye Motor (SEM) scale is used to assess children's responses during local anesthesia. Three parameters are considered: sound, eyes and motor skills. Each parameter is divided into 4 categories: comfort, mild comfort, moderate discomfort and severe discomfort, with corresponding scores from 1 to 4. The total score is derived by adding up the scores from these parameters, with a maximum possible score of 12 and a minimum of 3. A higher score is a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent university hospital, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patini R, Staderini E, Cantiani M, Camodeca A, Guglielmi F, Gallenzi P. Dental anaesthesia for children - effects of a computer-controlled delivery system on pain and heart rate: a randomised clinical trial. Br J Oral Maxillofac Surg. 2018 Oct;56(8):744-749. doi: 10.1016/j.bjoms.2018.08.006. Epub 2018 Aug 22. PMID 30143396